CLINICAL TRIAL: NCT03236467
Title: Neurobiological and Psychological Benefits of Exercise in Fibromyalgia and PTSD
Brief Title: Neurohormonal Benefits of Exercise in Fibromyalgia and PTSD
Acronym: EXFMPTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2395-P; 1I21RX002395-01A1 (NIH)
Record Dates: First submitted 2017-07-27; First posted 2017-08-02 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: FM and PTSD
Keywords: Fibromyalgia and PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Using an innovative translational research approach to study whether a 12 week-progressive - exercise program will reduce FM pain in patients with PTSD and to elucidate and modify potential PTSD-related deficiencies in neurobiological and psychological responses to exercise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FM + PTSD (Experimental): Individuals suffering from Fibromyalgia and PTSD
  Interventions: Behavioral: Progressive Exercise Training

INTERVENTIONS:
Behavioral: Progressive Exercise Training — Designed to ease primarily sedentary individuals into exercise training, increasing in intensity up to 80% of maximum Heart Rate Range over time.

SUMMARY:
The most recent conflicts are creating a new generation of Veterans, including an increasing number of women Veterans, who present with comorbid PTSD and chronic pain conditions, including Fibromyalgia (FM), from deployment-related physical injuries and exposure to psychological trauma. Health behavior change is important in treating these conditions and proactively preventing long-term negative health sequelae, in order to benefit these Veterans directly and reduce the challenges to our healthcare system. The proposed SPiRE application will use an innovative translational research approach to study whether a progressive -based exercise program will reduce FM pain in patients with PTSD and to elucidate and modify potential PTSD-related deficiencies in neurobiological and psychological responses to exercise to optimize the physical and psychological benefits of exercise for these individuals.

DETAILED DESCRIPTION:
Due to the COVID-19 pandemic, and after consultation with the appropriate research oversight, this study is temporarily suspended as of 3/15/20.

This study will compare the effects of a 12-week progressive exercise training program on 1) Fibromyalgia (FM) pain and PTSD symptoms, 2) pain threshold and tolerance, and 3) relevant biomarkers and neuromodulators including: a) anti-stress, anti-nociceptive, immune modulating factors such as neuropeptide Y (NPY) and GABAergic neuroactive steroids such as allopregnanolone and pregnanolone (together termed ALLO) b) factors that upregulate the expression of NPY and the GABAergic neuroactive steroids, and otherwise modulate inflammation, such as cortisol, c) excitatory factors such as substance P that directly promote pain transduction and d) pro-inflammatory cytokines such as IL-6 and IL-8 that not only increase pain and inflammation, but also contribute to psychological dysfunction (e.g. anhedonia and depression) via impact on the CNS reward system. This study will focus on Veterans with FM/PTSD. The study design includes a baseline, acute, cardiopulmonary exercise assessment (CPX) that will inform the exercise prescription for a 12-week "progressive exercise" training program, comprised of three 30-45 minute exercise sessions per week (walking or running, depending on the ability/capacity of the participant). Exercise sessions will be initially supervised by an exercise physiologist in the Clinical Studies Unit (CSU) at the VA Boston Healthcare System and then each participant will transition into the home. Weekly telephone calls by the PI will provide additional motivational support and problem solving. Implementation of the prescribed exercise regimen will also be supported by the use of heart rate and actigraph monitors programmed for the participant to achieve their prescribed heart rate range (HRR). Finally, an "endpoint" CPX assessment will occur at week 13 to track changes in psychological and neurobiological factors and to delineate their impact on pain and PTSD symptoms. Both CPX, maximum load, exercise tests will be performed in accordance with guidelines published by the American College of Cardiology. Among Veterans with FM/PTSD, changes in the biomarkers assessed after acute, CPX exercise testing will be associated with improvements in pain and PTSD symptoms.

Once identified, such biomarkers could be augmented by modification of the exercise regimen to help enhance the anti-stress hormone levels for the FM/PTSD population and experience clinically significant reductions in their symptoms. To obtain sufficient power, 36 participants (18/year) will be recruited. Data from this pilot work will be used to demonstrate feasibility and inform the further development of individually prescribed exercise regimens and a motivationally based exercise behavior change intervention aimed at reducing chronic musculoskeletal pain, including FM, and PTSD symptoms in Veterans. In the short-term, this SPiRE proposal will allow the PI to develop a more effective, motivationally based, exercise behavior change protocol that fosters long-term exercise adherence in patients with FM/PTSD. In the long-term, this intervention will be used as an adjunct to cognitive interventions for these disorders to be further developed and studied via a larger VA, NIH, or DOD-funded grant for which the PI will apply year 2 of the current SPiRE proposal.

ELIGIBILITY:
Inclusion Criteria:

* Only Veteran and civilian participants in whom a physical examination and medical history indicate that the participant meets current diagnostic criteria for FM, as specified by the American College of Rheumatology, will be eligible for the study.
* Eligible participants who agree to a blood draw for measurement of biomarkers, must be free of medications and other substances (e.g., illicit drugs and alcohol) that may alter results for 2-6 weeks depending on the medication and frequency of use (which must be cleared by MD consultants).
* If on pain medications with short half-lives, participants must be off of them for 5 half-lives before testing, generally about 24 hours.
* Any FM participant with an ICD-10 chronic pain diagnosis of a musculoskeletal etiology, will also be eligible for inclusion in the study as many individuals with FM also have such conditions.
* Any participant with a confirmed psychiatric diagnosis of PTSD will be included in the study. Individuals in the PTSD group must meet diagnostic criteria for current chronic PTSD (>3 months) as assessed by the CAPS-5, 1-Month Diagnostic Version.

Exclusion Criteria:

* Participants will be excluded from participation in the study if they have a life threatening or acute physical illness (e.g., cancer)
* Current schizophreniform illnesses (except for Psychosis NOS due to PTSD-related sensory hallucinations)
* Untreated bipolar disorder
* Or active suicidal or homicidal ideation requiring clinical intervention
* Individuals with current or past alcohol and/or substance dependence (less than three months from date of screening assessment) will be excluded
* Individuals seeking interventional pain treatment, such as surgical interventions or other pain clinic interventions, will also be excluded unless they agree to participate in the biomarker procedure prior to the start of their pain intervention.
* Finally, participants who have a neuropathic origin to their pain will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire-Revised | Two Years
  The FIQR has been found to be a useful and brief instrument to assess the overall impact and severity of FM.
  The FIQR consists of 21-items that assess pain, fatigue, stiffness, sleep, depression, memory, anxiety, balance, and environment sensitivity.
  All items are framed in the past 7 days and are scored on an 11-point numeric rating scores of 0 to 10.
  The total score ranges from 0 to 100, with higher scores representing greater symptom burden and functional limitations.

SECONDARY OUTCOMES:
Clinician Administered PTSD Scale -5 | Two Years
  This 30-item structured interview is designed to assess both the 17 symptoms of PTSD and the 8 hypothesized associated features. The scale yields a dichotomous diagnosis of PTSD, and also provides a continuous score of frequency and severity for each symptom. In addition, a behaviorally anchored probe question is provided for each symptom to increase the reliability of administration. The CAPS-5 is currently in the process of being validated however its previous version demonstrated excellent sensitivity (.81) and specificity (.95).57

CONTACTS AND LOCATIONS:
Overall Officials: Erica R. Scioli, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
This is a VABHS single site study. There are no plans to share the data outside of the VA Boston Healthcare System, unless specifically requested by authorized officials of VA.